CLINICAL TRIAL: NCT03974126
Title: Postprandial Effect of High-starch Meals in Individuals With Low and High Copy Number of the Salivary Amylase Gene
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: Dnr 2018/968
Record Dates: First submitted 2019-05-24; First posted 2019-06-04 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Postprandial Glucose and Insulin Response

STUDY DESIGN:
Intervention Model Description: Participants with low and high copy numbers of AMY1 were randomized to either 40 or 80 grams of starch in a crossover design.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Genotype were blinded for the participants and all research staff except for the principal investigator. Amount of bread was not blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 40 grams of starch to low and high AMY1 copy number carriers (Experimental): The postprandial response between individuals that are either carriers of low AMY1 copy numbers (2-4) or high copy numbers (10 or more copies) will be compared
  Interventions: Other: 40 grams of starch
- 80 grams of starch to low and high AMY1 copy number carriers (Experimental): The postprandial response between individuals that are either carriers of low AMY1 copy numbers (2-4) or high copy numbers (10 or more copies) will be compared
  Interventions: Other: 80 grams of starch

INTERVENTIONS:
Other: 40 grams of starch — 40 grams of starch in form of white bread to be consumed within 15 minutes
  Arms: 40 grams of starch to low and high AMY1 copy number carriers
Other: 80 grams of starch — 80 grams of starch in form of white bread to be consumed within 15 minutes
  Arms: 80 grams of starch to low and high AMY1 copy number carriers

SUMMARY:
Individuals with low copy numbers of salivary amylase gene have lower salivary amylase levels and might therefore have decreased capacity to metabolize starch into glucose. We will in a randomized crossover meal study examine the postprandial response of high-starch meals in individuals with either low or high copy number of the salivary amylase gene.

ELIGIBILITY:
Inclusion Criteria:

* Participant in the Malmö Offspring Study
* Genotyped for AMY1 copy number variation and selected for having either low (2-4) or high (10 or above) copy number of AMY1
* Gender: both males and females
* Completed information on dietary habits

Exclusion Criteria:

* Allergic to wheat, gluten intolerant or on a low-carbohydrate diet
* Inability to eat up to 4 slices of white bread in 15 minutes
* Use of medication known to influence glucose metabolism, appetite or saliva flow
* Diagnosed diabetes or high fasting plasma glucose (above 6.1 mmol/L)
* Smoking

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2019-09-19 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Postprandial glucose | AUC (0, 7, 15, 30, 45, 60, 90, 120 minutes)
  Postprandial glucose concentration assessed as incremental area under curve over 120 minutes (0, 7, 15, 30, 45, 60 ,90, 120 minutes)
Postprandial insulin | AUC (0, 7, 15, 30, 45, 60, 90, 120 minutes)
  postprandial insulin concentration assessed as incremental area under curve over 120 minutes (0, 7, 15, 30, 45, 60 ,90, 120 minutes)
Preabsorptive insulin release | 7 minutes
  Insulin concentration at 7 minutes

SECONDARY OUTCOMES:
subjective satiety | 0, 15, 30, 45, 60, 90, 120 minutes
  Visual analog scales (VAS) to evaluate hunger and satiety
salivary amylase activity | 0 minutes
  Salivary amylase activity will be measured by ELISA kits

OTHER OUTCOMES:
weight | 0 minutes
  weight will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- Lund University, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Farrell M, Ramne S, Gouinguenet P, Brunkwall L, Ericson U, Raben A, Nilsson PM, Orho-Melander M, Granfeldt Y, Tovar J, Sonestedt E. Effect of AMY1 copy number variation and various doses of starch intake on glucose homeostasis: data from a cross-sectional observational study and a crossover meal study. Genes Nutr. 2021 Nov 17;16(1):21. doi: 10.1186/s12263-021-00701-8. PMID 34789141